CLINICAL TRIAL: NCT01169090
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo Controlled Phase 2 Dose Finding Study Comparing the Safety, Tolerance, and Efficacy of Various Doses of SK-0403 Versus Placebo and Sitagliptin 100 mg in Patients Not Well-Controlled on Metformin Therapy
Brief Title: A Study Comparing the Safety, Tolerance, and Efficacy of Various Doses of SK-0403 Versus Placebo and Sitagliptin 100 mg in Patients Not Well-Controlled on Metformin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Roger Morgan, MD Chief Medical Officer, Kowa Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK-0403-2.01US
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SK-0403 100 mg QD (Experimental)
  Interventions: Drug: SK-0403
- SK-0403 200 mg QD (Experimental)
  Interventions: Drug: SK-0403
- SK-0403 400 mg QD (Experimental)
  Interventions: Drug: SK-0403
- SK-0403 200 mg BID (Experimental)
  Interventions: Drug: SK-0403
- Placebo (Sham Comparator)
  Interventions: Drug: Placebo
- Sitagliptin 100 mg QD (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: SK-0403 — SK-0403
  Arms: SK-0403 100 mg QD; SK-0403 200 mg BID; SK-0403 200 mg QD; SK-0403 400 mg QD
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Sitagliptin — Sitagliptin
  Arms: Sitagliptin 100 mg QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a range of doses of SK-0403 in subjects with type 2 diabetes that are not adequately controlled on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with type 2 diabetes between 18 and 75 years of age, inclusive
* Screening HbA1c between 7.0% to 10.0% for metformin stable subjects, 6.5% to 9.0% for subjects on metformin and 1 other antidiabetic agent (excluding thiazolidinediones, insulin, or incretin therapies [DPP-4 inhibitors and GLP-1 analogues]), or 7.5% to 11.0% for subjects on no antidiabetic medication or, if taking metformin, not on a stable dose of 1500 mg/day or maximum tolerated dose.
* No antidiabetic medication other than metformin for 3 months prior to randomization.
* Fasting plasma glucose less than 270 mg/dL (15 mmol/L) at screening.
* Body mass index between 20 kg/m2 and 45 kg/m2 inclusive at screening.

Exclusion Criteria:

* History of type 1 diabetes.
* Received treatment with insulin within 30 days of the screening visit or for more than 1 week within 3 months of the screening visit.
* Use of 3 or more oral antidiabetic medications at the time of the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to Week 16. | Baseline, 16 weeks
  Change in HbA1c from baseline to Week 16 with last observation carried forward (LOCF).

SECONDARY OUTCOMES:
Change from baseline in Fasting Plasma Glucose (FPG) | Baseline, 16 weeks

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Encinitas, California
  - Huntington Park, California
  - Los Angeles, California
  - San Mateo, California
  - Spring Valley, California
  - Walnut Creek, California
  - Miami, Florida
  - Palm Harbour, Florida
  - Pembroke Pines, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Paducah, Kentucky
  - New Orleans, Louisiana
  - Saint Paul, Minnesota
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Mount Giliad, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Charleston, South Carolina
  - Greensboro, South Carolina
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia